CLINICAL TRIAL: NCT04636372
Title: Effect of Meibomian Gland Related Therapy on the Morphology of Meibomian Gland
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: An one-month follow-up was completed after the treatment.
Sponsor: Yune Zhao (Other)
Responsible Party: Sponsor-Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LXY-meibomian gland
Record Dates: First submitted 2020-09-30; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-09

CONDITIONS: Xerophthalmia
MeSH Terms: conditions — Xerophthalmia | interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intense pulsed light therapy group (Experimental)
  Interventions: Device: Intense pulsed light therapy
- Hot compress massage group (Experimental)
  Interventions: Other: Hot compress massage
- Intense pulsed light therapy and hot compress massage group (Experimental)
  Interventions: Device: Intense pulsed light therapy; Other: Hot compress massage

INTERVENTIONS:
Device: Intense pulsed light therapy — Patients with xerophthalmia were treated with intense pulsed light of meibomian gland.
  Arms: Intense pulsed light therapy and hot compress massage group; Intense pulsed light therapy group
Other: Hot compress massage — Patients with xerophthalmia were treated with hot compress massage of meibomian gland.
  Arms: Hot compress massage group; Intense pulsed light therapy and hot compress massage group

SUMMARY:
200 participants at Eye Hospital of Wenzhou Medical University during September, 2020 to November, 2020 will be enrolled in this study. The meibomian gland related therapy are pulsed light therapy and meibomian gland hot compress massage.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with xerophthalmia

Exclusion Criteria:

* No history of ocular surgery and trauma
* Any eye diseases except xerophthalmia
* No treated for xerophthalmia before
* Successful completion of follow-ups

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
The length of meibomian glands after the treatment. | up to 2 months
  Length in millimeters.
The area of meibomian glands after the treatment. | up to 2 months
  Area in millimeters^2.
The percentage of meibomian glands after the treatment. | up to 2 months
  Percentage of meibomian glands in %(area of meibomian glands (mm^2) and area of palpebral conjunctiva (mm^2) will be combined to report percentage of meibomian glands in %) are used to assess this outcome measure.

IPD SHARING:
Plan to Share IPD: Undecided